CLINICAL TRIAL: NCT03309033
Title: Long-Term Immunologic Follow-Up of Women Who Received One, Two, and Three Doses of the Bivalent HPV Vaccine in the Costa Rica HPV-16/18 Vaccine Trial (CVT): Generating Durability Data: The ESCUDDO-CVT Study
Brief Title: Extended Follow-up of Women Who Received One, Two, and Three Doses of the HPV Vaccine in the Costa Rica Vaccine Trial (CVT), ESCUDDO-CVT Study
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCI-2020-07430; NCI-2020-07430 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20G012-07; 999917173; CEC-ICIC-E095-2017 (Other: National Cancer Institute)
Record Dates: First submitted 2017-10-12; First posted 2017-10-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Human Papillomavirus Infection; Human Papillomavirus-Related Malignant Neoplasm
MeSH Terms: conditions — Papillomavirus Infections | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire, biospecimen collection): Patients complete a short questionnaire regarding risk factors for HPV infection and undergo collection of blood samples for testing HPV16 and HPV18 levels on study.
  Interventions: Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This study is extending follow up of women who participated in the Costa Rica Vaccine Trial (CVT) and received one dose or two doses of the human papillomavirus (HPV) vaccine, along with a group of women who received three doses. It also studies the stability of HPV defenses in these groups of women for up to 20 years after initial vaccination. Studying samples of blood in the laboratory may provide information on how long one, two, and three doses of the vaccine provide protection against HPV. The results of this study may also help researchers learn whether one dose of HPV vaccine is enough to protect against HPV.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the change in antibody levels between years 11 and 20. II. Estimate the proportion of individuals who become seronegative (i.e.: serorevert) between years 11 and 20.

SECONDARY OBJECTIVES:

I. Assess the prevalence and distribution of type-specific HPV infections at least 18 years after HPV vaccination.

II. Assess the number and type of premalignant lesions present at least 18 years after vaccination.

III. For each dose regimen, characterize HPV-specific memory B cells and long-lived plasma cells present at least 18 years after HPV vaccination, and compare these characteristics with results from earlier time points.

OUTLINE: This is an observational study.

Patients complete a short questionnaire regarding risk factors for HPV infection and undergo collection of blood samples for testing HPV16 and HPV18 levels on study.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the CVT Long Term Follow-Up (LTFU) study

Exclusion Criteria:

* A random subset of the three-dose women

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women who participated in the Costa Rica Vaccine Trial and received the HPV vaccine
Sampling Method: Non-Probability Sample
Enrollment: 991 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Seropositivity | Up to 20 years after initial vaccination
  Negative/positive status will be assessed using the standard predefined cutoffs established at the testing laboratory.
Change in antibody levels | Between years 11 and 20 after initial vaccination
  Will report the geometric mean titer levels and their 95% confidence intervals at years 1, 2, 3, 4, 7, 9, 11, 14, 16, 18, and 20 for the 1-dose, 2-dose and 3-dose groups and for both human papillomavirus (HPV)-16 and HPV-18 antibodies. Will estimate these quantities using a weighted linear mixed models with log-titer level as the dependent variable and year as the independent variable, adjusting for laboratory batch and including a random-effects for participant and, when needed, participant: study year. For the three-dose analysis, will also include a covariate for study group. Moreover, will model the 19-year trend (e.g. excluding peak titers at year 1) by including time as a single continuous variable (i.e. linear effect) and then model time flexibly using a natural spline to assess a potentially non-linear relationship.
Proportion of individuals who serorevert | Between years 11 and 20 after initial vaccination
  For each dose regimen and for HPV 16, HPV 18, and a composite endpoint of either HPV type, will estimate the proportion of individuals who serorevert (i.e., become antibody negative by the assay cutoff) in years 1, 2, 3, 4, 7, 9, 11, 14, 16, 18, and 20. Will also report 95% confidence intervals for these estimates. Again, will follow the approach described in our previous work. Note, will consider both standard and updated cutoffs and will use batch-adjusted levels. Can obtain the relative risk for seroreversion and its 95% confidence interval using score tests. Will then use generalized linear mixed models with seroreversion as the outcome and all other parameters similar to above to assess trends over time.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee R Kreimer, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Agencia Costarricense de Investigaciones Biomédicas (ACIB), Liberia, Guanacaste Province, Costa Rica